CLINICAL TRIAL: NCT07228806
Title: Evaluation of the Effectiveness of Telerehabilitation on Pelvic Floor Dysfunction in Postpartum Women: A Single-Blind Randomised Controlled Trial
Brief Title: Effectiveness of Telerehabilitation on Pelvic Floor Dysfunction at Postpartum Woman
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Naz Kalem, PM&R Specialist, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AEŞH-EK-2025-062
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Postpartum Pelvic Floor Function and Symptoms
Keywords: Postpartum Woman; Pelvic Floor Dysfunction; Telerehabilitation
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental)
  Interventions: Other: Pelvic floor exercises with telerehabilitation
- Conventional group (Active Comparator)
  Interventions: Other: Pelvic floor exercises without telerehabilitation

INTERVENTIONS:
Other: Pelvic floor exercises with telerehabilitation — Patients in the telerehabilitation group will be assigned the same 8-week exercise programme as those in the conventional group to be carried out at home. Unlike the conventional group, patients in the telerehabilitation group will be contacted by telephone each week throughout the exercise programme to check their adherence to the programme, to ask if they have encountered any problems with the exercise programme, and to answer any questions they may have.
  Arms: Telerehabilitation group
Other: Pelvic floor exercises without telerehabilitation — An 8-week exercise programme consisting of 45-minute Kegel exercises and core stabilisation exercises per day will be provided for implementation at home in the conventional group.
  Arms: Conventional group

SUMMARY:
These events are largely due to pelvic floor dysfunction that develops after pregnancy. Kegel exercises and core stabilisation exercises performed in the postpartum period are important in preventing pelvic floor dysfunction. However, considering the mother's adaptation process to both the baby and her new life in the postpartum period, there may be problems with exercise compliance. Increasing exercise compliance through telerehabilitation can be effective in preventing pelvic floor dysfunction and improving women's quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 45
2. Primiparous women
3. Term vaginal delivery
4. 6 weeks postpartum
5. Willingness to participate in the study

Exclusion Criteria:

1. Presence of faecal or urinary incontinence prior to pregnancy
2. Use of assisted delivery devices (vacuum, forceps)
3. Presence of neurological disease
4. Presence of psychiatric illness or cognitive problems that make it difficult to answer questions
5. Caesarean section delivery
6. History of diabetes mellitus
7. Perineal rupture

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor muscle strength assessment | Before exercises programme and 8th week of exercises programme
  Pelvic floor muscle strength assessment using the SineBravo 2-channel EMG Biofeedback device

SECONDARY OUTCOMES:
Measurement of the distance between the inferior edge of the pubic symphysis and the anteromedial edge of the puborectalis muscle using transperineal ultrasound | Before exercises programme and 8th week of exercises programme
Pelvic floor questionnaire for pregnant and postpartum women | Before exercises programme and 8th week of exercises programme
Female Sexual Function Index | Before exercises programme and 8th week of exercises programme

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)